CLINICAL TRIAL: NCT01988675
Title: MRI Study of Radiation-Induced Damage to White Matter and Blood-Brain-Barrier
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2003.083; HUM00040138 (Other: University of Michigan)
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms | interventions — Neuropsychological Tests; Magnetic Resonance Imaging; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Partial Brain Irradiation: Patients will receive partial brain irradiation for malignant or benign brain tumors as standard of care. Patients will also have MRI (Magnetic Resonance Imaging) scans and neuropsychological/QOL (Quality of Life Questionnaire) tests prior during and after RT (Radiation Therapy).
  Interventions: Radiation: Partial Brain Irradiation; Behavioral: Neuropsychological Testing; Behavioral: Quality of Life Questionnaire; Device: Magnetic Resonance Imaging (MRI) Assessments
- Whole Brain Irradiation: Patients will receive whole brain irradiation for brain metastases as standard of care. Patients will also have MRI (Magnetic Resonance Imaging) scans and neuropsychological/QOL (Quality of Life Questionnaire) tests prior during and after RT (Radiation Therapy).
  Interventions: Radiation: Whole Brain Irradiation; Behavioral: Neuropsychological Testing; Behavioral: Quality of Life Questionnaire; Device: Magnetic Resonance Imaging (MRI) Assessments

INTERVENTIONS:
Radiation: Whole Brain Irradiation
  Groups: Whole Brain Irradiation
Radiation: Partial Brain Irradiation
  Groups: Partial Brain Irradiation
Behavioral: Neuropsychological Testing
Behavioral: Quality of Life Questionnaire
Device: Magnetic Resonance Imaging (MRI) Assessments — MRI Assessments include Diffusion Tensor Imaging (DTI)and Gd-DTPA (Diethylenetriamine Pentaacetic Acid - a radioactive tracer injected into the patient and viewed on images).

SUMMARY:
This is a study to determine if Magnetic Resonance Imaging (MRI) techniques can detect early changes in white matter (in the brain) and the blood-brain barrier resulting from radiation therapy.

DETAILED DESCRIPTION:
Patients will be assigned to one of two groups based on the type of radiation they will be receiving: whole brain irradiation or partial brain irradiation. Patients will undergo Magnetic Resonance Imaging (MRI) assessments, neurocognitive testing (Quality of Life and Neuropsychological assessments), and clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving partial brain irradiation for malignant or benign brain tumors (including low-grade gliomas, high-grade gliomas, malignant meningioma, pituitary adenomas, supratentorial meningioma, or craniopharyngiomas); or patients receiving whole brain irradiation for brain metastases.
* Patients must be 18 years of age or older
* Patients must sign a study specific consent form approved by the Institutional Review Board (IRB) of the University of Michigan prior to study entry.
* Patients must have a neurological function class 1 or 2 with a Karnofsky performance status (a scoring system used to quantify general well being and quality of life on a scale of 100 to 0) of greater than or equal to 70.
* Patients must have an expected life expectancy of greater than 6 months.

Exclusion Criteria:

* Patients with a history of major medical illness or psychiatric impairment which, in the investigator's opinion, will prevent administration of the protocol.
* Patients who have had prior external beam irradiation to the brain or head/neck area that will lead to overlap of the radiation field.
* Patients should have no contraindications to having a contrast enhanced Magnetic Resonance Imaging (MRI) scan.
* Prisoners are excluded.
* Pregnant women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving partial or whole brain radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2004-08-26 (Actual); Primary Completion 2014-06-03 (Actual); Study Completion 2014-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Magnetic Resonance Imagining (MRI) with different radiation dose at different timepoints. | Baseline, at 3 weeks on radiation therapy (RT) (partial brain irradiation only), last week of RT, 6 weeks post RT, 4 months post RT (whole brain irradiation only), 6 months post RT, 18 months post RT (partial brain irradiation only)
  Linear mixed models will be used to relate Magnetic Resonance Imagining (MRI) changes and radiation dose.

SECONDARY OUTCOMES:
Associate changes in Magnetic Resonance Imagining (MRI) assessments with changes in neurocognitive function and clinical symptoms, from baseline, and at different timepoints. | Baseline, 6 weeks post radiation therapy (RT), 4 months post RT (whole brain irradiation only), 6 months post RT, 18 months post RT (partial brain irradiation only)
  Changes in Magnetic Resonance Imagining (MRI) assessments will be compared graphically to changes in neurocognitive function and clinical symptoms. Parallel analysis will be conducted on each of the neurocognitive tests to determine if MRI assessments can identify patients at increased risk for later neurocognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Cao, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hosptial, Ann Arbor, Michigan, United States